CLINICAL TRIAL: NCT00336167
Title: Clinical Trial on the Effect of Bezafibrate in the Muscular Form of Carnitine Palmitoyltransferase 2 Deficiency
Brief Title: Bezafibrate Trial in CPT2 Deficiency
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Association Française contre les Myopathies (AFM), Paris (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-05-19
Record Dates: First submitted 2006-06-09; First posted 2006-06-13 (Estimated); Last update posted 2007-04-09 (Estimated); Status verified 2007-04

CONDITIONS: Carnitine Palmitoyl Transferase 2 Deficiency
Keywords: carnitine palmitoyl transferase 2 deficiency; Fatty acid oxidation; Mitochondria
MeSH Terms: conditions — Carnitine palmitoyl transferase 2 deficiency | interventions — Bezafibrate; Pharmaceutical Preparations

INTERVENTIONS:
Drug: bezafibrate (drug)

SUMMARY:
The purpose of this study is to determine whether bezafibrate is effective in the treatment of the muscular adult form of carnitine palmitoyltransferase 2 deficiency

DETAILED DESCRIPTION:
Fatty acids are the main source of energy for non-glucodependent tissues during fasting and prolonged exercise. Carnitine Palmitoyltransferase (CPT) 1 and 2 are a key-enzymes in the regulation of mitochondrial FAO, by governing entry of long-chain fatty acids within the mitochondrial matrix. CPT2 deficiency is among the most common inherited disorders of mitochondrial fatty acid oxidation (FAO). The neonatal and infantile forms of CPT2 deficiency are life-threatening diseases with a hepatocardiomuscular presentation. The adult form presents as recurrent attacks of rhabdomyolysis, mostly triggered by prolonged exercise, fasting, and infections, and is usually considered as a "mild" disease. However, patients commonly suffers permanent muscle weakness, and/or frequent (weekly, and sometimes daily) attacks of rhabdomyolysis, that occasionally result in severe episodes of acute renal insufficiency, and rarely in sudden death.

Difference in the clinical severity of the distinct forms of CPT2 deficiency correlates in some extent with in vitro data. Thus, when measured in fibroblasts or lymphocytes, the residual CPT2 activity and the long-chain fatty acid oxidation (LCFAO) are usually less than 10% of control values in the neonatal and infantile forms, while they most often are over 20 % of controls in the adult form.

Clinical management of CPT2-deficient patients remains poor, and most often does not succeed in significantly improving their clinical condition. Treatment mostly relies so far on restriction in lipid intake and limitation of fasting and exercise. We decided a few years ago to set up a project of pharmacological therapy for this disease, based upon in vitro testing of pharmacological agents potentially able to increase the residual enzymatic activity in CPT2-deficient cell lines. Some of the best "candidate" drugs were PPAR agonists, used since over two decades as hypolipidemic drugs. PPAR alpha is a transcription factor belonging to the superfamily of steroid-thyroid nuclear receptors, that has been shown to regulate the constitutive expression of the CPT2 gene and protein in the adult mouse heart and liver and to mediate up-regulation of the CPT2 gene in response to fibrates in mouse liver. We recently shown that bezafibrate, a PPAR alpha agonist, was able to restore close to the normal the apparent CPT2 activity and the LCFAO in both fibroblasts and cultured myoblasts from several patients with the adult form of CPT2 deficiency. Therefore, the purpose of the current application is to test in vivo the potentially beneficial effect of bezafibrate therapy in a cohort of 12 patients with the adult form of this disease. All patients are clinically managed by either of the 2 research groups involved in this project, namely the Neurology department of l'hospital Pitié-Salpétrière and the Genetics department of l'hospital Necker-Enfants Malades. Patients fulfilling inclusion criteria will first be submitted to a 6-month period of clinical and biological survey, with a written registration of each clinical symptoms, and measurement of CK activity once a month. The initial examination will include i) muscular testing, ii) measurement of CPT2 activity , LCFAO, and quantitation of CPT2 transcripts both in lymphocytes and in a fresh small sample of skeletal muscle, and iii)assay of acylcarnitines, a compound accumulated upstream of the metabolic block, in blood. Bezafibrate will thereafter be daily supplied as a 400 to 600 mg dose, according to the renal function, for 6 months. Follow-up will focus on the muscular symptomatology and on the hepatic, muscular, and renal tolerance of the treatment. At the end of the clinical trial, each patient will be submitted to an examination similar to the initial one, including a second muscle biopsy used for measurement of CPT2 activity , LCFAO, and amount of CPT2 transcripts. It has to be emphasized that, for the first time, such a therapy should impact directly the cause of the disease (the defective enzyme activity) and not only its consequences (accumulation of cell lipid and defective energy production).

ELIGIBILITY:
Inclusion Criteria:

* occurrence of at least 5 attacks of rhabdomyolysis or of severe myalgias per year, AND/OR permanent muscle weakness objectivized by muscle testing outside a rhabdomyolysis attack AND
* significant decrease in both the CPT2 activity and the rate of long-chain fatty acid oxidation measured in lymphocytes and/or in a skeletal muscle sample outside a rhabdomyolysis attack

Exclusion Criteria:

* age below 18 years
* less than 5 attacks of rhabdomyolysis or severe myalgias per year AND absence of muscle impairment detected by muscle testing
* liver failure, renal failure, hyperhomocysteinemia prior to setting up the bezafibrate therapy
* treatment with another hypolipidemic drug ("statins) or with anticoagulant
* pregnancy or lactation during the period of fibrate therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2006-06; Study Completion 2007-07 (Estimated)

PRIMARY OUTCOMES:
Rate of 3H-palmitate oxidation in the patients'lymphocytes and skeletal muscle

SECONDARY OUTCOMES:
Rate of CPT2 enzymatic activity in the patients'lymphocytes and skeletal muscle
Rate of palmitoyl-L-carnitine oxidation in the patients' skeletal muscle
Steady-state amount of CPT2 mRNA in the patients'skeletal muscle

CONTACTS AND LOCATIONS:
Overall Officials: Bruno EYMARD, M.D, Study Chair — Service de Neurologie 2 Groupe hospitalier Pitié-Salpétriere, Paris, France; Jean Paul BONNEFONT, M.D., Ph D,, Principal Investigator — Unite INSERM U781
Locations (1):
- Jean Paul Bonnefont, Paris, France